CLINICAL TRIAL: NCT03745742
Title: Post Myocardial Infarction's Rehabilitation Guided by Heart Rate Variability
Acronym: HRV REEDUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Clinique cardio-pneumologique de Durtol (Unknown); Almerys (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-417; 2015-AO1755-44 (Other: 2015-AO1755-44)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Myocardial Infarction; Cardiac Rehabilitation
Keywords: Cardiac rehabilitation; myocardial infarction; heart rate variability; physical fitness
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Other): standard rehabilitation protocol according to the personal functional capacities (measured by a cardiopulmonary test on the beginning of the cardiac reeducation.
  Interventions: Other: HRV measurement
- study strategy (Experimental): individualization of the rehabilitation program according to the daily HRV measure and the personal functional capacity (measured by a cardiopulmonary test on the program beginning).
  Interventions: Other: HRV measurement

INTERVENTIONS:
Other: HRV measurement — Patients in group A (control) will benefit from a standard re-training protocol based on initial functional abilities. The training is done at a target heart rate corresponding to the heart rate reached at the first ventilatory threshold (about 55% of VO2max).
  * Patients in group B (study strategy) will benefit from a re-training protocol based on HRV and initial functional abilities. Any increase in HRV compared to the previous day will result in an increase in workload of 10Watt. Any increase or decrease in HRV for 3 days in a row will cause the stagnation of the workload for 2 days.
  HRV is measured every day in each group via a heart rate belt and a smartphone App.
  Other Names: Rehabilitation program based on HRV measurement

SUMMARY:
Cardiac rehabilitation reduces morbidity and mortality after myocardial infarction (MI) and improve the sympathovagal balance. The autonomic nervous system (ANS) can be explored by the variation of heart rate (HRV). The HRV is a fatigue marker and guides the athletes training programs. A smartphone app can measure the HRV via a heart rate monitor.

The main study objective is to compare the effect on the functional capacities of a re-training adapted to the HRV compared to a standard program in the post-MI The secondary objective is to compare the patients' quality of life according to the rehabilitation program and to validate the HRV smartphone app.

This is a prospective, multicenter study. Post-MI patients treated with angioplasty with a LVEF> 40% are randomized into 2 groups: HRV (re-training adapted to HRV daily: 10W decrease or increase in workload according to the HRV) or control (continuous training in SV1). Patients underwent a cardiopulmonary test, a walking test (TM6) and a SF36 questionaries' at the entrance and exit. The taking of HRV was done every morning in a standardized way via the smartphone app during the 20 re-training sessions.

DETAILED DESCRIPTION:
Description of the study:

Patients with myocardial infarction (STEMI or NSTEMI) without alteration of left ventricle systolic function, agreeing to participate at a cardiac rehabilitation program will be included in the study and randomized into two groups:

* Group A (= control): standard rehabilitation protocol according to the personal functional capacities (measured by a cardiopulmonary test on the beginning of the cardiac reeducation.)
* Group B (= strategy to the study): individualization of the rehabilitation program according to the daily HRV measure and the personal functional capacity (measured by a cardiopulmonary test on the program beginning).

The duration of the rehabilitation program will be 4 weeks with 5 training sessions per week (Monday to Friday), or 20 training sessions. At the end of the program, patients will benefit from an assessment of functional abilities and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Man, Woman ≥18 years old and <70 years old
* STEMI or NSTEMI having undergone angioplasty revascularization at least 8 day before the beginning of reeducation
* Sinus rhythm
* LVEF> 40% (Simpson Biplane echocardiography

Exclusion Criteria:

* Contraindications to cardiac re-training:
* Ventricular or supraventricular rhythm disorder
* Heart failure.
* Pericardial effusion.
* STEMI or NSTEMI <J8
* NSTEMI or STEMI , post revascularization by bypass surgery
* Non-sinus rhythm
* Comorbidity preventing all sports activity: severe AOMI; amputation; neurological disorder, hemiplegia.
* Pathology leading to modifications of the HRV:
* Chronic lung disease
* Renal insufficiency with clearance <30 ml / min (MDRD)
* LVEF <40%
* Electrical cardiac stimulation
* Linked to the person:
* Protected Majors
* People unable to express their consent.
* Pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
gain of VO2max | after 4 weeks of cardiac rehabilitation
  The gain obtained after 4 weeks of cardiac rehabilitation(expressed as% basal value) of VO2max

SECONDARY OUTCOMES:
patients'quality of life after 4 weeks of cardiac rehabilitation | after 4 weeks of cardiac rehabilitation
  The taking of HRV was done every morning in a standardized way via the smartphone app during the 20 re-training sessions.
The patient's functional capacity after 4 weeks of cardiac rehabilitation estimated by the distance covered during the 6-minute walk test. | after 4 weeks of cardiac rehabilitation
  The gain in meter at the 6 minutes' walk test

CONTACTS AND LOCATIONS:
Overall Officials: D'Agrosa Boiteux Marie-Claire, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France